CLINICAL TRIAL: NCT06139055
Title: A 2-part, Phase 1, Randomized Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Comparative Bioavailability of Multiple-ascending Doses of GSBR-1290 in Healthy Overweight/Obese Participants
Brief Title: A Study of Multiple-ascending Doses of GSBR-1290 in Healthy Overweight/Obese Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSBR-1290-05
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Capsules; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is open-label, 2-period, 2-sequence, cross-over and Part 2 is double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 (Sequence 1: Capsule to Tablet): GSBR-1290 Capsule/GSBR-1290 Tablet (Experimental): Participants will receive a single dose of GSBR-1290 oral capsule formulation on Day 1 in Treatment Period 1 followed by GSBR-1290 oral tablet formulation on Day 8 (Day 1 of Treatment Period 2).
  Interventions: Drug: GSBR-1290 (Capsule/Tablet)
- Part 1(Sequence 2: Tablet to Capsule): GSBR-1290 Tablet/GSBR-1290 Capsule (Experimental): Participants will receive a single dose of GSBR-1290 oral tablet formulation on Day 1 in Treatment Period 1 followed by GSBR-1290 oral capsule formulation on Day 8 (Day 1 of Treatment Period 2).
  Interventions: Drug: GSBR-1290 (Capsule/Tablet)
- Part 2 (Cohort 1): GSBR-1290/Placebo Tablet (Experimental): Participants will receive GSBR-1290 or matching-placebo oral tablets once daily for a total of 12 weeks.
  Interventions: Drug: GSBR-1290; Drug: Placebo
- Part 2 (Cohort 2): GSBR-1290/Placebo Tablet (Experimental): Participants will receive GSBR-1290 or matching-placebo oral tablets once daily for a total of 12 weeks.
  Interventions: Drug: GSBR-1290; Drug: Placebo
- Part 2 (Cohort 3): GSBR-1290/Placebo Tablet and GSBR-1290/Placebo Capsule (Experimental): Participants will receive GSBR-1290 or matching-placebo oral tablets once daily for a total of 12 weeks. In the last 4 weeks, participants will be further randomized to GSBR-1290 capsules or tablets or matching-placebo at Week 9 to 10 followed by alternate (capsule or tablet) formulation of either GSBR-1290 or placebo at Week 11 to 12.
  Interventions: Drug: GSBR-1290 (Capsule/Tablet); Drug: Placebo (Capsule/Tablet)

INTERVENTIONS:
Drug: GSBR-1290 (Capsule/Tablet) — Participants will receive GSBR-1290 oral capsules or tablets.
  Arms: Part 1 (Sequence 1: Capsule to Tablet): GSBR-1290 Capsule/GSBR-1290 Tablet; Part 1(Sequence 2: Tablet to Capsule): GSBR-1290 Tablet/GSBR-1290 Capsule; Part 2 (Cohort 3): GSBR-1290/Placebo Tablet and GSBR-1290/Placebo Capsule
Drug: GSBR-1290 — Participants will receive GSBR-1290 oral tablets.
  Arms: Part 2 (Cohort 1): GSBR-1290/Placebo Tablet; Part 2 (Cohort 2): GSBR-1290/Placebo Tablet
Drug: Placebo — Participants will receive matching-placebo oral tablets.
  Arms: Part 2 (Cohort 1): GSBR-1290/Placebo Tablet; Part 2 (Cohort 2): GSBR-1290/Placebo Tablet
Drug: Placebo (Capsule/Tablet) — Participants will receive matching-placebo oral capsules or tablets.
  Arms: Part 2 (Cohort 3): GSBR-1290/Placebo Tablet and GSBR-1290/Placebo Capsule

SUMMARY:
The purpose of this study is to compare the safety, tolerability, pharmacokinetic (PK), and comparative bioavailability of repeated administration of GSBR-1290 in healthy overweight/obese participants.

DETAILED DESCRIPTION:
This is a 2-part study in which Part 1 will compare the PK of GSBR-1290, administered as tablet and capsule, using a 2-period, 2-sequence, crossover design in approximately 16 healthy overweight/obese participants. Part 2 will evaluate multiple-ascending doses of GSBR-1290 tablet in 3 cohorts, using 3 different titration regimens. Secondly in Part 2, the study will evaluate the comparative bioavailability of GSBR-1290 tablet versus capsule at a potentially clinically efficacious dose at steady state in Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

1. Provided evidence of a signed informed consent before any study-related activities are initiated and be willing to comply with all study procedures.
2. Healthy overweight or obese adult men and women.
3. Age greater then or equal to (>=)18 and less than or equal to (<=) 75 years.
4. Body mass index (BMI) >=27.0 kilogram per square meter (kg/m^2).

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurological disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Part 1: Analysis of Maximum Observed Plasma Concentration (Cmax) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate Pharmacokinetic (PK) Parameters | From start of study drug up to Day 10
Part 1: Analysis of Time to Maximum Observed Plasma Concentration (Tmax) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 10
Part 1: Analysis of Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 10
Part 1: Analysis of Area Under the Plasma Concentration-time Curve From 0 to infinity (AUC0-inf) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 10
Part 1: Analysis of Apparent Terminal Elimination Half-life (t1/2) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 10
Part 1: Analysis of Total Apparent Body Clearance (CL/F) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 10
Part 1: Analysis of Apparent Volume of Distribution (Vz/F) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 10
Part 2: Number of Participants With Adverse Events (AEs) and Serious AEs | From start of study drug up to End of study (EOS) in Part 2 (up to Day 98)
Part 2: Number of Participants With Severity of AEs | From start of study drug up to EOS in Part 2 (up to Day 98)
Part 2: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | From start of study drug up to EOS in Part 2 (up to Day 98)
Part 2: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters | From start of study drug up to EOS in Part 2 (up to Day 98)
Part 2: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters | From start of study drug up to EOS in Part 2 (up to Day 98)

SECONDARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AEs) and Serious AEs | From start of study drug up to EOS in Part 1 (Day 17)
Part 1: Number of Participants Based on Severity of AEs | From start of study drug up to EOS in Part 1 (Day 17)
Part 1: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to EOS in Part 1 (Day 17)
Part 1: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters | Baseline up to EOS in Part 1 (Day 17)
Part 1: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters | Baseline up to EOS in Part 1 (Day 17)
Part 2: Analysis of Maximum Observed Plasma Concentration (Cmax) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate Pharmacokinetic (PK) Parameters | From start of study drug up to Day 84
Part 2: Analysis of Time to Maximum Observed Plasma Concentration (Tmax) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 84
Part 2: Analysis of Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval (24 hours) at Steady State (AUC0-tau) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 84
Part 2: Analysis of Plasma Trough Concentrations for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 84
Part 2: Analysis of Apparent Terminal Elimination Half-life (t1/2) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | From start of study drug up to Day 84

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - ERG Clinical (Clinical Pharmacology of Miami - CPMI), Miami, Florida
  - Syneos Miami Site, Miami, Florida
  - Parexel Baltimore Early Phase Clinical Unit, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product have been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Structure Therapeutics does not grant external requests for individual de-identified patient data for the following purposes:
  * re-evaluating safety and efficacy end points already addressed in the product labelling,
  * assessing safety or efficacy for an indication in current development
  Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.